CLINICAL TRIAL: NCT07084298
Title: Effects of 12 Weeks of Oral Iron Supplementation on Skeletal Muscle Iron Content, Mitochondrial Function, and Indices of Aerobic Fitness in Healthy Females With Suboptimal Iron Stores
Brief Title: Effects of Iron Supplementation on Skeletal Muscle Properties in Females With Suboptimal Iron Storage
Acronym: MyoIRON
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Martin MacInnis, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: REB25-0927
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Iron Deficiency
Keywords: iron; iron deficiency; athletic performance; female athlete; iron supplements; ferritin; hemoglobin; muscle; muscle ferritin; mitochondria; critical power; aerobic fitness; exercise; placebo
MeSH Terms: conditions — Iron Deficiencies; Motor Activity | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron supplement (Experimental): Dietary supplement: Oral iron supplement, encapsulated ferrous sulphate (150mg elemental iron)
  Interventions: Dietary Supplement: Oral iron supplement
- Placebo (Placebo Comparator): Placebo control: Sugar pill, encapsulated polysaccharide substance (malodextrin)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Oral iron supplement — Encapsulated ferrous sulphate (150mg elemental iron)
  Arms: Iron supplement
Other: Placebo — Encapsulated polysaccharide (maltodextrin)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn whether oral iron supplementation will increase skeletal muscle iron storage and its effects on exercise capacity in females with suboptimal iron status. The study will include healthy females, ages 18-40, who either have suboptimal or optimal iron stores.

The main questions it aims to answer are:

* Does iron supplementation increase skeletal muscle iron storage and alter the expression of iron-related and mitochondrial proteins?
* Does iron supplementation improve single-leg exercise performance?
* Is serum ferritin correlated with the abundance of iron-related proteins in skeletal muscle?

Researchers will compare outcomes from females with suboptimal iron status who receive oral iron supplementation to those who receive a placebo to see if supplementation improves muscle iron storage, protein expression, and exercise performance. Additionally, a non-intervention control group with optimal iron status will be included to assess baseline differences.

Participants will:

- Be randomly assigned to receive 150 mg elemental iron or placebo (maltodextrin) every other day for 12 weeks

Complete pre- and post-supplementation testing, including:

* Blood draws to assess iron status
* Skeletal muscle biopsies to analyze protein content
* Whole-body and single-leg exercise tests to assess performance
* Controls will undergo baseline-only testing to compare physiological and biochemical markers

DETAILED DESCRIPTION:
This study is intended to evaluate the effects of oral iron supplementation on muscle iron levels in females with suboptimal iron status. The design involves both a randomized controlled trial (RCT) for those with low blood iron levels, as well as a cross-sectional component, including only healthy controls. Iron supplementation will be administered to half of those enrolled in the RCT portion to evaluate the effects of iron uptake within the muscle. Therefore, the primary goal of the study is to determine if iron is stored within the muscle in meaningful amounts following an extended period of oral iron supplementation in healthy females with suboptimal iron status.

The study's rationale extends from the high prevalence of low iron levels among females globally, especially among those who are involved in endurance sports. At the level of the muscle, iron serves in several key biological functions, including oxygen transport, energy production, and even recovery from exercise, making it essential for performance. Although the investigators understand some amount of iron is stored within the muscle, the investigators are currently unaware whether meaningful changes occur following a period of supplementation. Therefore, the proposed protocol outlined below is designed to test the hypothesis that taking iron for a prolonged period at adequate doses will result in meaningful changes.

Participants involved in this study will include biological females aged 18-40 with suboptimal iron status (blood ferritin ≤50 µg/L), who are otherwise healthy, for the RCT portion, or normal iron status (blood ferritin ≥50 µg/L) for healthy controls. Interested participants will be screened, and those eligible for the RCT will be randomly assigned to either an oral iron supplement or a placebo sugar pill, ensuring that the encapsulation is preserved to promote blinding. Participants will consume the assigned treatment once every 2nd day for 12 weeks. Exercise and other biological tests will be performed both before and after supplementation during the RCT, while healthy controls will only participate in baseline testing.

The following is an overview of the study design:

Baseline testing

This phase involves five visits and approximately 6.5 hours of laboratory testing spread over two weeks. Participants in the RCT and those acting as healthy controls will both complete the baseline testing phase.

Visit I: Blood draw

Participants will report to the laboratory in the fasted condition. They will be verbally informed of the methods of this study by the researcher and given time to ask questions before their written consent is obtained. Participants will complete a short survey to characterize their menstrual cycle. Subsequently, an individual trained in phlebotomy will collect venous blood for analysis from an antecubital vein using appropriate techniques. Following analysis of the blood iron markers, participants will be informed whether they are eligible to participate in the RCT or serve as a control. This visit will take approximately 1 hour.

Visit II: Body composition scan and familiarization

Participants will arrive fasted and undergo a body composition scan via dual-energy x-ray absorptiometry (DXA), which takes approximately 10 minutes. They will then be permitted to eat and drink. Participants will complete additional questionnaires (to be repeated before each exercise testing session) detailing perceived rest and food records. They will then be familiarized with a dynamic knee extension (i.e., kicking) task involving 15 minutes of exercise at varying intensities with feedback on technique. Once familiarized, participants will perform a single-leg incremental ramp protocol to determine their quadriceps peak power. In this test, participants will kick at a fixed cadence (e.g., 40 kicks per minute) while resistance gradually increases until they are unable to continue due to fatigue or personal choice. This test will last approximately 10 to 20 minutes. This visit will take approximately 1.5 hours.

Visit III: V̇O₂max and familiarization

On a separate day, at least 24 hours after the last visit, participants will return to the lab without fasting. They will complete an incremental ramp exercise test on a cycle ergometer (double-leg) to measure V̇O₂max, characterizing their aerobic fitness. This test involves gradually increasing resistance until the participant can no longer continue. After a rest period of at least 20 minutes (or longer if needed), participants will perform additional familiarization with the dynamic knee extension exercise, consisting of 30 minutes of kicking at various intensities. This visit will take approximately 1.5 hours.

Visit IV: Lower-body power, quadriceps oxidative capacity, and critical power

On a separate day, at least 24 hours after their last visit, participants will return to the lab without fasting. During this visit, participants will perform countermovement jumps and undergo testing of quadriceps oxidative capacity (OxCap) and critical power (CP) in their dominant leg. They will begin with OxCap testing, which involves a brief isometric contraction of the knee extensor muscles followed by repeated short arterial occlusions using a rapid cuff inflator. This test is performed in duplicate. Next, participants will perform countermovement jumps - a series of vertical jumps on a force plate repeated three times with 60-second rests in between. After resting for 10 to 15 minutes, they will perform three bouts of dynamic knee extension at different intensities to task failure to determine CP. Each bout will last 2 to 20 minutes and be separated by at least 20 minutes of rest. This visit will take approximately 2 hours.

Visit V: Muscle biopsy procedure

On a separate day, at least 24 hours after their last visit, participants will return to the lab in a fasted state for a muscle biopsy. A physician will obtain a small muscle sample using the proper technique, which will later be analyzed for iron-related and mitochondrial protein content. This visit will take approximately 45 minutes.

Supplementation phase

This phase involves two visits and approximately one hour of laboratory testing. Only participants in the RCT will complete this phase.

Participants in the RCT will be randomized to receive either an iron supplement or a placebo in a 1:1 ratio using a concealed allotment procedure. Participants will consume either one iron pill (150 mg elemental iron) or one placebo pill (PolyCal, maltodextrin) every other day for 12 weeks. Each iron supplement contains 50 mg of elemental iron, while the placebo includes none. This dosing protocol is based on prior research showing that alternate-day dosing improves gastrointestinal tolerance. Both iron and placebo pills will be encapsulated within a gelatin capsule for blinding, ensuring no difference in release rate.

Visits VI and VII: Week 4 and 8 blood draws

Participants will visit the lab during weeks 4 and 8 of their supplementation period to provide blood samples. Before each blood draw, they will complete questionnaires about gastrointestinal symptoms and a food record covering the previous three days. Blood will be collected by a trained individual using a standard venipuncture technique. Each visit will take approximately 30 minutes.

Post-supplementation testing

Post-supplementation testing will involve the same procedures as baseline testing, but the visits will be slightly more condensed and re-ordered. In total, participants will visit the lab three times over approximately two weeks for about 5.5 hours of testing. Only RCT participants will complete this phase.

Visit VIII: Blood draw, muscle biopsy, and body composition scan.

After completing supplementation, participants will return to the lab in a fasted state to provide a blood sample and a muscle biopsy, and to undergo a body composition scan. Participants will also repeat familiarization with the single-leg exercise task, using the same procedure from visit II. They will complete questionnaires on gastrointestinal symptoms and their three-day food record. This visit will take approximately 2 hours.

Visits IX and X: Exercise testing

These visits are identical to visits III and IV from the baseline phase and will take the same amount of time (1.5 and 2 hours, respectively) over approximately one week. They will begin a minimum of 48 hours after visit VIII and be separated by at least 24 hours. Before each test, participants will complete questionnaires about rest and their food records for the preceding three days. After all testing is complete, participants and researchers will record their guess about which supplement was consumed to assess the effectiveness of blinding. Participants will then be informed of their group allocation.

ELIGIBILITY:
Inclusion Criteria:

* biologically female
* between the ages of 18-40 years of age at the time of enrolment
* plasma ferritin ≤ 50 µg/ L (RCT) or >50 µg/L (controls)
* complete Get Active Questionnaire (GAQ: Canadian Society for Exercise Physiology) without contraindication

Exclusion Criteria:

* have a body mass index (BMI) > 30 kg/m2
* taking medications that have been shown to affect cardiovascular, respiratory, or metabolic responses to exercise (e.g., β-blockers, anti-inflammatories, anti-coagulants, insulin, etc.)
* hemoglobin ≤ 120 g/L (anemia cut-off for women)
* have known health problems or contraindications that prohibit exercise, including renal or gastrointestinal disorders, metabolic disease, heart disease, vascular disease, arthritis, diabetes, respiratory disease, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions that are being treated and deemed likely to confound the results
* dieting for weight loss or following a low-carbohydrate diet (known to affect iron homeostasis)
* history of smoking or using tobacco products
* consuming excessive amounts of alcohol (>21 units/week)
* supplementing with iron (>5mg/day) in the last 3 months
* any blood donation or surgeries in the past 3 months
* antibiotic use within the previous four weeks before study enrolment
* current laxative use
* known history of thalassemia
* known bleeding disorder
* chronic use of nonsteroidal anti-inflammatory drugs
* Currently/last 3 months taking prescription medications that are known to affect iron absorption (i.e. Antacids/PPIs (e.g., omeprazole), H2 Blockers (e.g., ranitidine), Tetracycline Antibiotics (e.g., doxycycline), Quinolone Antibiotics (e.g., ciprofloxacin), Cholestyramine, Colchicine, Methyldopa).
* currently pregnant or plans to get pregnant within the duration of the study, and
* do not understand English
* Participants will be removed from the study if they begin taking any other forms of supplemental iron or choose to donate blood

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Muscle Ferritin | At baseline (week 0) and completion of supplementation (week 12)
  Muscle collection: The muscle biopsy involves the removal of a small piece of muscle tissue from the vastus lateralis using a sterile hollow needle. The area over the incision site will be carefully cleaned, and a small amount of local anesthetic will be injected into and under the skin. A small, 4 - 5 mm incision will be made in the skin to create an opening for the biopsy needle.
  The biopsy needle will then be inserted through the incision into the muscle, and a small piece of muscle (~50 mg) will be removed, and the needle taken out. A medical doctor will perform this procedure.
  Protein analysis: Western blotting will be used to analyze the abundance of ferritin within small sections of the muscle sample.

SECONDARY OUTCOMES:
Serum iron status | Every four weeks beginning at baseline (week 0) until completion of supplementation (week 12)
  A forearm venous blood draw (10ml): Samples will be sent to a third-party laboratory for analysis of blood biomarkers, including ferritin and hemoglobin.
Iron-related proteins | At baseline (week 0) and completion of supplementation (week 12)
  Muscle collection: The muscle biopsy involves the removal of a small piece of muscle tissue from the vastus lateralis using a sterile hollow needle. The area over the incision site will be carefully cleaned, and a small amount of local anesthetic will be injected into and under the skin. A small, 4 - 5 mm incision will be made in the skin to create an opening for the biopsy needle.
  The biopsy needle will then be inserted through the incision into the muscle, and a small piece of muscle (~50 mg) will be removed, and the needle taken out. A medical doctor will perform this procedure.
  Protein analysis: Small sections of each muscle sample will undergo Western blotting to analyze other iron-related proteins (e.g., transporters)
Mitochondrial proteins | At baseline (week 0) and completion of supplementation (week 12)
  Muscle collection: The muscle biopsy involves the removal of a small piece of muscle tissue from the vastus lateralis using a sterile hollow needle. The area over the incision site will be carefully cleaned, and a small amount of local anesthetic will be injected into and under the skin. A small, 4 - 5 mm incision will be made in the skin to create an opening for the biopsy needle.
  The biopsy needle will then be inserted through the incision into the muscle, and a small piece of muscle (~50 mg) will be removed, and the needle taken out. A medical doctor will perform this procedure.
  Protein analysis: Small sections of each muscle sample will undergo Western blotting to analyze potential changes to mitochondrial protein content (e.g., transporters). Other sections of the same sample will undergo enzyme assays to quantify the relative changes in protein activity within the sample.
Whole body aerobic fitness (VO2max) | At baseline (week 0) and completion of supplementation (week 12)
  Exercise: Participants will complete an incremental ramp exercise test on a cycle ergometer (double-leg) to measure V̇O2max, serving to characterize participants' aerobic fitness. For this test, participants will cycle on a stationary bicycle while the resistance increases gradually until the participants are unable to continue because they are fatigued and/or wish to stop (~10-20 min)
  Metabolic analysis: For whole-body exercise tests, participants will wear a face mask attached to a metabolic cart (Quark CPET, COSMED, Rome, Italy) that will analyze the volume and content of expired breath to determine oxygen uptake, carbon dioxide production, and minute ventilation. The maximal whole-body rate of oxygen consumption (V̇O2max) will be determined as the highest 30s average from a ramp incremental test.
Single-leg critical power | At baseline (week 0) and completion of supplementaton (week 12)
  Exercise: Participants will perform three bouts of dynamic knee extension exercise at differing intensities to task failure to determine their CP. Each bout of kicking will last between 2 and 20 minutes and be separated by a minimum of 20 minutes of rest.
  Critical power determination: The two parameters of the intensity-duration relationship, CP (W) and W' (J), will be calculated using three equations: the linear work-time model, the inverse linear model, and the hyperbolic model.
  Linear work-time model: W = CP × t + W' Inverse linear model: P = W' × (1/t) + CP Hyperbolic model: t = W' / (P - CP)
  Where P represents power output and W represents the total work completed. The equation with the highest coefficient of determination (R2) and lowest standard error of the estimate will be selected to determine CP and W' for each participant.
Muscle oxidative capacity | At baseline (week 0) and completion of supplementation (week 12)
  Exercise: Participants will complete oxidative capacity testing, which involves performing a brief isometric contraction of the knee extensor muscles followed by repeated, transient (5 s) arterial occlusions with a rapid cuff inflator. This protocol will be performed in duplicate.
  Oxidative measure: Near-infrared spectroscopy (NIRS) will be used to non-invasively measure muscle oxidative capacity. The NIRS device will be held in place with two-sided tape and a tensor bandage on the vastus lateralis muscle, and a blood pressure cuff will be wrapped around the upper portion of the thigh, proximal to the NIRS device. During transient (5 s) arterial occlusions following a brief exercise stimulus, NIRS will be used to measure changes in the concentration of oxygenated and deoxygenated hemoglobin. Using these measures, the rate at which muscle oxygen uptake recovers following a series of brief contractions, a surrogate for the oxidative capacity of the muscle, can be determined.
Countermovement jump test | At baseline (week 0) and completion of supplementation (week 12)
  Exercise: Participants will perform a countermovement jump that involves completing a series of short-burst vertical jumps on a force plate to assess lower-body power and explosiveness. This activity will be repeated twice more, separated by 60 s of rest, before resting for several (~10-15) mins.

CONTACTS AND LOCATIONS:
Overall Officials: Martin J MacInnis, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rineau E, Gueguen N, Procaccio V, Genevieve F, Reynier P, Henrion D, Lasocki S. Iron Deficiency without Anemia Decreases Physical Endurance and Mitochondrial Complex I Activity of Oxidative Skeletal Muscle in the Mouse. Nutrients. 2021 Mar 24;13(4):1056. doi: 10.3390/nu13041056. PMID 33805065
- [Background] Paul BT, Manz DH, Torti FM, Torti SV. Mitochondria and Iron: current questions. Expert Rev Hematol. 2017 Jan;10(1):65-79. doi: 10.1080/17474086.2016.1268047. Epub 2016 Dec 12. PMID 27911100
- [Background] Ohira Y, Hegenauer J, Strause L, Chen CS, Saltman P, Beinert H. Mitochondrial NADH dehydrogenase in iron-deficient and iron-repleted rat muscle: an EPR and work performance study. Br J Haematol. 1982 Dec;52(4):623-30. doi: 10.1111/j.1365-2141.1982.tb03938.x. PMID 6291576
- [Background] Moretti D, Goede JS, Zeder C, Jiskra M, Chatzinakou V, Tjalsma H, Melse-Boonstra A, Brittenham G, Swinkels DW, Zimmermann MB. Oral iron supplements increase hepcidin and decrease iron absorption from daily or twice-daily doses in iron-depleted young women. Blood. 2015 Oct 22;126(17):1981-9. doi: 10.1182/blood-2015-05-642223. Epub 2015 Aug 19. PMID 26289639
- [Background] MacInnis MJ, Zacharewicz E, Martin BJ, Haikalis ME, Skelly LE, Tarnopolsky MA, Murphy RM, Gibala MJ. Superior mitochondrial adaptations in human skeletal muscle after interval compared to continuous single-leg cycling matched for total work. J Physiol. 2017 May 1;595(9):2955-2968. doi: 10.1113/JP272570. Epub 2016 Aug 3. PMID 27396440
- [Background] Jacobs A. Tissue changes in iron deficiency. Br J Haematol. 1969 Jan-Feb;16(1):1-4. doi: 10.1111/j.1365-2141.1969.tb00372.x. No abstract available. PMID 5795211
- [Background] Hinton PS, Giordano C, Brownlie T, Haas JD. Iron supplementation improves endurance after training in iron-depleted, nonanemic women. J Appl Physiol (1985). 2000 Mar;88(3):1103-11. doi: 10.1152/jappl.2000.88.3.1103. PMID 10710409
- [Background] Frise MC, Holdsworth DA, Johnson AW, Chung YJ, Curtis MK, Cox PJ, Clarke K, Tyler DJ, Roberts DJ, Ratcliffe PJ, Dorrington KL, Robbins PA. Abnormal whole-body energy metabolism in iron-deficient humans despite preserved skeletal muscle oxidative phosphorylation. Sci Rep. 2022 Jan 19;12(1):998. doi: 10.1038/s41598-021-03968-4. PMID 35046429
- [Background] DellaValle DM, Haas JD. Iron supplementation improves energetic efficiency in iron-depleted female rowers. Med Sci Sports Exerc. 2014 Jun;46(6):1204-15. doi: 10.1249/MSS.0000000000000208. PMID 24195864
- [Background] Stugiewicz M, Tkaczyszyn M, Kasztura M, Banasiak W, Ponikowski P, Jankowska EA. The influence of iron deficiency on the functioning of skeletal muscles: experimental evidence and clinical implications. Eur J Heart Fail. 2016 Jul;18(7):762-73. doi: 10.1002/ejhf.467. Epub 2016 Jan 21. PMID 26800032
- [Background] Newhouse IJ, Clement DB, Taunton JE, McKenzie DC. The effects of prelatent/latent iron deficiency on physical work capacity. Med Sci Sports Exerc. 1989 Jun;21(3):263-8. PMID 2733574
- [Background] Melenovsky V, Hlavata K, Sedivy P, Dezortova M, Borlaug BA, Petrak J, Kautzner J, Hajek M. Skeletal Muscle Abnormalities and Iron Deficiency in Chronic Heart FailureAn Exercise 31P Magnetic Resonance Spectroscopy Study of Calf Muscle. Circ Heart Fail. 2018 Sep;11(9):e004800. doi: 10.1161/CIRCHEARTFAILURE.117.004800. PMID 30354361
- [Background] McDougall RM, Tripp TR, Frankish BP, Doyle-Baker PK, Lun V, Wiley JP, Aboodarda SJ, MacInnis MJ. The influence of skeletal muscle mitochondria and sex on critical torque and performance fatiguability in humans. J Physiol. 2023 Dec;601(23):5295-5316. doi: 10.1113/JP284958. Epub 2023 Oct 30. PMID 37902588
- [Background] Hinton PS. Iron and the endurance athlete. Appl Physiol Nutr Metab. 2014 Sep;39(9):1012-8. doi: 10.1139/apnm-2014-0147. Epub 2014 May 27. PMID 25017111
- [Background] Finch CA, Miller LR, Inamdar AR, Person R, Seiler K, Mackler B. Iron deficiency in the rat. Physiological and biochemical studies of muscle dysfunction. J Clin Invest. 1976 Aug;58(2):447-53. doi: 10.1172/JCI108489. PMID 956378
- [Background] Dietz JV, Fox JL, Khalimonchuk O. Down the Iron Path: Mitochondrial Iron Homeostasis and Beyond. Cells. 2021 Aug 25;10(9):2198. doi: 10.3390/cells10092198. PMID 34571846
- [Background] Dallman PR, Beutler E, Finch CA. Effects of iron deficiency exclusive of anaemia. Br J Haematol. 1978 Oct;40(2):179-84. doi: 10.1111/j.1365-2141.1978.tb03655.x. No abstract available. PMID 361066
- [Background] Caswell AM, Tripp TR, Kontro H, Edgett BA, Wiley JP, Lun V, MacInnis MJ. The influence of sex, hemoglobin mass, and skeletal muscle characteristics on cycling critical power. J Appl Physiol (1985). 2024 Jul 1;137(1):10-22. doi: 10.1152/japplphysiol.00120.2024. Epub 2024 May 23. PMID 38779761
- [Background] Brownlie T 4th, Utermohlen V, Hinton PS, Giordano C, Haas JD. Marginal iron deficiency without anemia impairs aerobic adaptation among previously untrained women. Am J Clin Nutr. 2002 Apr;75(4):734-42. doi: 10.1093/ajcn/75.4.734. PMID 11916761
- [Background] Brutsaert TD, Hernandez-Cordero S, Rivera J, Viola T, Hughes G, Haas JD. Iron supplementation improves progressive fatigue resistance during dynamic knee extensor exercise in iron-depleted, nonanemic women. Am J Clin Nutr. 2003 Feb;77(2):441-8. doi: 10.1093/ajcn/77.2.441. PMID 12540406